CLINICAL TRIAL: NCT01829191
Title: Controlling Myopia Progression With Soft Contact Lenses
Brief Title: Controlling Myopia Progression With Soft Contact Lenses (Contact Lens Control)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-1561AD
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Results first posted 2015-07-29 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Lens A (Experimental): Test lenses will be worn in a daily wear modality
  Interventions: Device: Soft Contact Test Lens A
- Test Lens C (Experimental): Test lenses will be worn in a daily wear modality
  Interventions: Device: Soft Contact Test Lens C

INTERVENTIONS:
Device: Soft Contact Test Lens A — FDA-approved, non-marketed daily disposable soft contact lens, conventional design
  Arms: Test Lens A
Device: Soft Contact Test Lens C — Daily disposable soft contact lens with new optical design
  Arms: Test Lens C

SUMMARY:
This study is to investigate whether novel soft contact lens optical designs can slow myopia progression

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be between 8 and 12 years of age.
2. At least one of the subject's parents or legal guardian must read and understand English or Chinese.
3. The subject's manifest objective refraction (measured with an auto refractor) must be sphere: between -0.25D and -4.50D, and cylinder: <1.50D in each eye.
4. The subject's best sphere contact lens correction must lie between -0.75D (better of the two eyes)and -4.25D (poorer of the two eyes).
5. The subject's cycloplegic objective refraction must be here: between -0.75D and -4.00D cylinder: < or equal to 1.00D in each eye.
6. The subject must have 1.00D or less difference in spherical equivalent between the two eyes with cycloplegic refraction.
7. The subject must have a spectacle lens best-corrected visual acuity of 0.8 (20/25) or better in both eyes.
8. The subject's parent or legal guardian must read and sign the STAEMENT OF INFORMED CONSENT and the subject must read and sign the Child's Assent Form and be provided a copy of each form.
9. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.

Exclusion Criteria:

1. Ocular or systemic allergies or diseases that may interfere with contact lens wear.
2. Systemic disease or autoimmune disease or use of medications (e.g. antihistamine), which may interfere with contact lens wear.
3. Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormality of the cornea, which may contraindicate contact lens wear.
4. Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection that might interfere with contact lens wear.
5. Any ocular infection.
6. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
7. Any infectious disease (e.g. hepatitis, tuberculosis) or an immunosuppressive disease (e.g. HIV)
8. Diabetes
9. Anisometropia of greater than 1.00D by cycloplegic refraction.
10. Astigmatism of greater than 1.00D in either eye by cycloplegic refraction.
11. Eye injury or surgery within eight weeks immediately prior to enrollment for this study.
12. Previous refractive surgery, orthokeratology, keratoconus, or other corneal irregularity in either eye. Rigid contact lens wearers cannot be enrolled in the study unless they are off rigid contact lenses for at least 4 weeks.
13. Strabismus in either eye.
14. Pupil or lid abnormality or infection in either eye
15. Central corneal scar in either eye
16. Aphakia in either eye
17. Contraindications to contact lens wear such as dry eye or history of prior unsuccessful contact lens wear.
18. History of participation in prior clinical trials aimed to control myopia progression.
19. Surgically altered eyes, ocular infection of any type, ocular inflammation.
20. An anterior chamber angle grade 2 or narrower by the Van Herrick method

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 174 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2010-05-01 (Actual); Study Completion 2010-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston, Massachusetts, United States

REFERENCES:
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645
- [Derived] Cheng X, Xu J, Brennan NA. Accommodation and its role in myopia progression and control with soft contact lenses. Ophthalmic Physiol Opt. 2019 May;39(3):162-171. doi: 10.1111/opo.12614. PMID 30994197

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of those 174 screened subjects, 42 were ineligible to participate in the study and 5 eligible subjects did not randomize to the study arm.
Groups:
- Test Lens C: Test lens will be worn in a daily wear modality
Period: Overall Study
Arm/Group | Test Lens A | Test Lens C
Started | 63 | 64
Completed | 56 | 50
Not Completed | 7 | 14
Not completed — Relocation | 0 | 1
Not completed — Lens discomfort | 0 | 3
Not completed — Lens handling difficulty | 1 | 4
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Subject was fit for ortho - k | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline summary was conducted on all subjects who randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Lens A | Test Lens C | Total
Number analyzed (Participants) | 63 | 64 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 63 | 64 | 127
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (1.1) | 9.7 (1.1) | 9.7 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 29 | 30 | 59
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 64 | 127

OUTCOME MEASURES:

1. Primary Outcome: Spherical Equivalent Refractive Error
Description: Cycloplegic spherical equivalent auto refraction of the subject's right eye was computed from the sphero-cylindrical refraction measured with an open-field auto refractor. The median of 3 repeated measures, each of which was the average of 3 consecutive readings, was used for the analysis. Higher values in spherical refraction indicate progression in Myopia.
Time Frame: Baseline and every 6 months post-baseline for 2 years
Population: Analysis was conducted on all randomized subjects who have at least one data point.
Measure: Mean (Standard Error); unit: diopter (D)
Arm/Group | Test Lens A | Test Lens C
Number analyzed (Participants) | 59 | 53
diopter (D)
  Change from baseline 6 months | -0.386 (0.3270) | -0.185 (0.2873)
  Change from baseline 12 months: number analyzed (Participants) | 57 | 52
  Change from baseline 12 months | -0.679 (0.5253) | -0.548 (0.4050)
  Change from baseline 18 months: number analyzed (Participants) | 24 | 16
  Change from baseline 18 months | -0.934 (0.4761) | -0.614 (0.4140)
  Change from baseline 24 months: number analyzed (Participants) | 13 | 11
  Change from baseline 24 months | -1.054 (0.4559) | -1.080 (0.6800)

2. Secondary Outcome: Axial Length
Description: Axial length was measured with the IOLMaster at baseline and every 6 months for 2 years. Five measurements were collected for each visit from the subject's right eye and the average of the five measurements was used for the analysis.
Time Frame: Baseline and every 6 months for 2 years
Population: Analysis was conducted on all randomized subjects who have at least one data point.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Test Lens A | Test Lens C
Number analyzed (Participants) | 59 | 53
millimeter (mm)
  Change from baseline 6 months | 0.172 (0.1029) | 0.061 (0.1038)
  Change from baseline 12 months: number analyzed (Participants) | 57 | 52
  Change from baseline 12 months | 0.371 (0.1471) | 0.229 (0.1581)
  Change from baseline 18 months: number analyzed (Participants) | 24 | 16
  Change from baseline 18 months | 0.479 (0.2049) | 0.313 (0.1946)
  Change from baseline 24 months: number analyzed (Participants) | 13 | 11
  Change from baseline 24 months | 0.545 (0.2177) | 0.514 (0.2808)

ADVERSE EVENTS:
Groups:
- All Subjects: All subjects who eligible to participate in the study whether or not randomized to the study arm.
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/132
Other Adverse Events (participants affected / at risk) | 0/132

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes